CLINICAL TRIAL: NCT00237224
Title: Open Label Study of Postmenopausal Women With ER and /or PgR Positive Breast Cancer Treated With Letrozole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345EMX01
Record Dates: First submitted 2005-10-09; First posted 2005-10-12 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer, ER and/or PgR positive, Letrozole
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

ARMS (1):
- FEM345 (Experimental)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole

SUMMARY:
To evaluate safety and efficacy (measured by clinical tumor response) of letrozole daily dose, 2.5 mg in postmenopausal patients with primary (untreated) breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal woman able to comply with the protocol requirements with primary invasive breast cancer, histologically confirmed by core needle biopsy, whose tumors are estrogen (ER) and / or progesterone (PgR) positive, defined by core biopsy immunohistochemistry with > 10% positive malignant epithelial cells.
2. Clinical stage *T2, T3, T4a,b,c, N0, 1 or 2, M0

   * Clinical stage T2 tumors which in the Investigators opinion would not be eligible for breast-conserving surgery.
3. Post menopausal status defined by one of the following:

   * No spontaneous menses for at least 1 year, in women > 55 years.
   * Spontaneous menses within the past 1 year but amenorrhoeic in women ≤ 55 years (e.g. spontaneous or secondary to hysterectomy), and with postmenopausal gonadotrophin levels (LH y FSH levels > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dl) or according to the definition of "postmenopausal range" for the laboratory involved.
   * Bilateral oophorectomy. (Prior to the diagnosis of breast cancer).
4. Tumor measurable by clinical examination, mammography and ultrasound.

Exclusion Criteria:

1. Prior treatment with letrozole or tamoxifen.
2. Uncontrolled endocrine disorders such as diabetes mellitus, confirmed hypo- or hyperthyroidism, Cushing's Syndrome, Addison's disease (treated or untreated).
3. Patients with unstable, angina, or uncontrolled cardiac disease (e.g. Class III or IV New York Heart association's Functional Classification).
4. Patients with bilateral breast tumors
5. Patients who are eligible for breast conserving surgery
6. Evidence of inflammatory breast cancer or distant metastasis.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-02; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Identify Eg and/or Pg receptors in breast cancer patients in adjuvant treatment with tamoxifen for 4-5 years | 4 months

SECONDARY OUTCOMES:
Identify the number of patients in adjuvant treatment with tamoxifen within 4-5 years or close to end this treatment time | 4 months
Determine the relation of positive Eg / Pg receptors vs negative (unknown) Eg / Pg receptors and the only selection criteria for the adjuvant treatment with tamoxifen is postmenopause status | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Guadalajara, Zacatecas, México DF, Mexico